CLINICAL TRIAL: NCT06866717
Title: Relative Effectiveness of a Hybrid Prehabilitation Program (Home-based and Center-based) Compared to a Center-based Prehabilitation Program Before Non-small Cell Lung Cancer Surgery: A Randomized Controlled Equivalence Study
Brief Title: Hybrid Prehabilitation Before Thoracic Surgery
Acronym: HYBREATH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ADIR Association (Other)
Collaborators: Région Normandie (Other Government); Département de la Seine Maritime (Unknown); European Union (Other); French-Speaking Association of Supportive Care in Cancer (AFSOS) (Unknown); MSD France (Industry); Union des Kinésithérapeutes Respiratoires (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HYBREATH
Record Dates: First submitted 2025-02-19; First posted 2025-03-10 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Prehabilitation; Telerehabilitation; Hybrid prehabilitation; Home-base exercise training
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Single-center, randomized controlled equivalence trial with concealed allocation, a blinded assessor, and an intention-to-treat analysis.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hybrid prehabilitation (Experimental): 15 prehabilitation sessions divided into 3 center-based sessions and 12 home-based sessions.
  Interventions: Other: Hybrid prehabilitation
- Centre-based prehabilitation. (Active Comparator): 15 center-based prehabilitation sessions.
  Interventions: Other: Center-based prehabilitation

INTERVENTIONS:
Other: Hybrid prehabilitation — Hybrid prehabilitation group (15 sessions in total over 3 weeks): participants will complete 3 center-based sessions and 12 home-based sessions over three weeks. The home-based sessions will mirror those in the center-based group (initiation, training session, final session).
  For the home-based component, participants will receive a cycle ergometer, pulse oximeter, activity tracker, and a tablet application for guidance throughout the program, remote monitoring and communication (TELEREHAPP). Home-based sessions include:
  * Endurance training on the cycle ergometer (15 to 45 minutes per session).
  * Strength training and balance exercises (30 minutes per session).
  * Inspiratory muscle training (10 sets of 10 repetitions at 30% of maximal inspiratory pressure).
  * Physical activity coaching with daily step count objective;
  * Regular remote monitoring and support via the tablet application, with weekly check-ins from healthcare professionals.
  Arms: Hybrid prehabilitation
Other: Center-based prehabilitation — Center-based prehabilitation group (15 sessions in total over 3 weeks): participants will attend 15 sessions in the center, over three weeks, comprising:
  * 1 initiation session (approximately 3 hours) including preoperative patient education, instructions on the use of inspiratory muscle training device, endurance training on a cycle ergometer, strength training, and balance exercises.
  * 13 endurance training sessions (1.5 to 2 hours each) focusing on endurance training (15 to 45 minutes), strength training (30 minutes), and inspiratory muscle training (10 sets of 10 repetitions at 30% of maximal inspiratory pressure).
  * 1 final session (2 to 2.5 hours) with a review of the program and educational reinforcement.
  Arms: Centre-based prehabilitation.

SUMMARY:
Background and study aims:

Lung cancer is a leading cause of cancer-related deaths worldwide. Patients with non-small cell lung cancer often undergo lung surgery to remove the tumor. Before surgery, patients may participate in prehabilitation programs to improve their physical fitness and overall health, which can lead to better surgical outcomes. Traditionally, these programs are conducted entirely in specialized centers, but places are scarce, limiting access. This study aims to compare the relative effectiveness of a hybrid prehabilitation program, combining home-based and center-based sessions, with the standard center-based program. The primary goal is to assess changes in aerobic capacity, measured by peak oxygen uptake, before and after participation in the prehabilitation program.

Who can participate?

Adults over 18 years old who are scheduled for lung resection surgery to treat diagnosed or suspected non-small cell lung cancer can participate. Participants should be referred for respiratory prehabilitation in a preoperative context and live at home with another adult, present during exercise sessions. The surgery date should be either not yet established at the time of inclusion or scheduled for at least four weeks later. Participants should have a peak oxygen uptake of less than 20 ml/kg/min, be beneficiaries of a social security system, and have read and understood the information letter and signed the consent form.

What does the study involve?

This is a single-center, randomized controlled trial with two groups:

Center-based prehabilitation group: Participants will attend 15 sessions over three weeks (five sessions per week) at the center. The program includes an initial session of therapeutic education and exercise training, followed by 13 prehabilitation sessions, and a final session with educational reinforcement.

Hybrid prehabilitation group: Participants will have three sessions at the center and 13 sessions at home over the same period. They will be provided with equipment such as a cycle ergometer, pulse oximeter, physical activity sensor, and a tablet application (TELEREHAPP) to guide and monitor their home-based exercises. Regular phone contact with healthcare professionals will be maintained for support.

All participants will undergo assessments before and after the program, including an incremental exercise test on a cycle ergometer to measure peak oxygen uptake.

What are the possible benefits and risks of participating?

Participants may experience improved physical fitness, which could lead to better surgical outcomes and reduced postoperative complications. The study will also provide insights into the relative effectiveness of hybrid prehabilitation, potentially offering more flexible options and facilitating access to care for future patients. Risks may include muscle soreness, fatigue, or injury related to exercise, independently of group allocation. All exercise sessions will be supervised or monitored to minimize these risks. Participants will receive instructions on how to perform exercises safely and will be encouraged to report any adverse effects promptly.

DETAILED DESCRIPTION:
Lung cancer is a leading cause of cancer-related mortality worldwide. Surgical resection is the primary curative treatment for early-stage non-small cell lung cancer; however, patients often present with compromised physical fitness, which can adversely affect surgical outcomes and postoperative recovery.

Prehabilitation, the process of enhancing a patient's functional capacity before surgery, has emerged as a promising strategy to improve surgical outcomes. Studies have demonstrated that prehabilitation can lead to reductions in postoperative complications, shorter hospital stays, and improved quality of life.

Prehabilitation programs are typically conducted in specialized clinical settings, which may limit accessibility and adherence. Hybrid models that combine home-based and center-based interventions may offer the opportunity for a more flexible option and may address the limited access to specialized care for many patients.

This study primarily aims to evaluate the relative effectiveness of a hybrid prehabilitation program of 15 sessions (incorporating both home-based and center-based components) compared to a center-based prehabilitation program of 15 sessions in patients undergoing surgery for non-small cell lung cancer on the change in oxygen uptake.

The study also aims to evaluate the relative effectiveness of a hybrid prehabilitation program of 15 sessions (incorporating both home-based and center-based components) compared to a center-based prehabilitation program of 15 sessions in patients undergoing surgery for non-small cell lung cancer on the change in peak power output, ventilatory efficiency, functional capacity, quadriceps muscle maximal isometric strength, respiratory muscle strength, maximal peak expiratory flow and cough expiratory flow, quality of life, psychological status as well as adherence, postoperative complications, clinically relevant postoperative complications, length of hospital stay, and environmental impact.

Study design:

This is a prospective, monocentric, randomized controlled equivalence trial with concealed allocation and a single-blind design (blinded evaluator). Participants will be randomly assigned to one of two groups:

Center-based prehabilitation group (15 sessions in total over 3 weeks): participants will attend 15 sessions in the center, over three weeks, comprising:

1 initiation session (approximately 3 hours) including preoperative patient education, instructions on the use of inspiratory muscle training device, endurance training on a cycle ergometer, strength training, and balance exercises.

13 endurance training sessions (1.5 to 2 hours each) focusing on endurance training (15 to 45 minutes), strength training (30 minutes), balance training, and inspiratory muscle training (10 sets of 10 repetitions at 30% of maximal inspiratory pressure).

1 final session (2 to 2.5 hours) with a review of the program and educational reinforcement.

Hybrid prehabilitation group (15 sessions in total over 3 weeks): participants will complete 3 center-based sessions and 12 home-based sessions over three weeks. The center-based sessions will mirror those in the center-based prehabilitation group (initiation, training session, final session). For the home-based component, participants will receive a cycle ergometer, pulse oximeter, activity tracker, and a tablet application (TELEREHAPP) for guidance throughout the program, remote monitoring, and communication. Home-based sessions include:

Endurance training on the cycle ergometer (15 to 45 minutes per session).

Strength training and balance exercises (30 minutes per session).

Inspiratory muscle training (10 sets of 10 repetitions at 30% of maximal inspiratory pressure).

Physical activity coaching, including a daily step goal.

Regular remote monitoring and support via the tablet application, with weekly check-ins from healthcare professionals.

Sample size calculation for equivalence study:

Assuming a mean change difference in peak oxygen uptake between the two groups of 0 ml/kg/min, a significance level (alpha) of 0.05, a power of 80%, an equivalence margin of 1.75 ml/kg/min, and a standard deviation of 1.8 ml/kg/min for the change in peak oxygen uptake after a condensed rehabilitation program of 5 sessions per week during 3 weeks, we plan to recruit 19 patients per group, totaling 38 patients.

Statistical analysis:

Categorical data will be presented as counts (percentages). Continuous descriptive data will be expressed as means (SD) or medians (IQR), depending on their distribution. The normality of distributions will be assessed using the Kolmogorov-Smirnov test.

Intergroup differences will be reported as mean differences (95% confidence intervals). Non-parametric data will be converted to means (SD) using an appropriate method. Results will be interpreted based on the span of the 95% confidence intervals relative to pre-specified outcomes (see Outcome Measures section).

The relative effect of interventions on categorical data will be examined using relative risk (95% confidence intervals).

Statistical analyses will be conducted on an intention-to-treat basis, using the last available observation for preoperative assessment criteria and considering the absence of complications for postoperative complications (for patients who will not ultimately be operated).

A secondary per-protocol analysis will be performed.

A sensitivity analysis will be conducted by including baseline values as a covariate in the model.

Analyses will be performed using GraphPad 8 and R software.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient scheduled to undergo lung resection for the treatment of diagnosed or suspected bronchial cancer
* Referred for prehabilitation before lung resection surgery
* Patient living at home with another adult present during exercise sessions
* Surgery date not established at the time of inclusion in the program, or at least 4 weeks away
* Peak oxygen uptake below 20 ml/kg/min
* Affiliated with a health insurance system
* Able to read and understand the information letter and sign the consent form

Non-Inclusion Criteria:

* Oxygen therapy during exercise
* Cardiological contraindication to exercise training
* Concomitant neoadjuvant chemoradiotherapy
* Refusal to participate in a center-based prehabilitation training program
* Orthopedic, neurological, vascular, or neuromuscular conditions limiting exercise training on a cycle ergometer
* Patient under guardianship or curatorship
* Pregnant or breastfeeding women

Exclusion Criteria:

-Withdrawal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in peak oxygen uptake. | From enrollment to the end of prehabilitation (15 sessions, 3 weeks).
  Change in peak oxygen uptake will be assessed during an incremental cardiopulmonary exercise testing on a cycle ergometer before and after the prehabilitation program. The pre-specified minimal clinically important difference is set at 1.75ml/kg/min.

SECONDARY OUTCOMES:
Change from baseline in peak power output. | From enrollment to the end of prehabilitation (15 sessions, 3 weeks).
  Change in peak power output will be assessed during an incremental cardiopulmonary exercise testing on a cycle ergometer before and after the prehabilitation program. The pre-specified minimal clinically important difference is set at 4 watts.
Change from baseline in ventilatory efficiency. | From enrollment to the end of prehabilitation (15 sessions, 3 weeks).
  Change in ventilatory efficiency will be assessed during an incremental cardiopulmonary exercise testing on a cycle ergometer before and after the prehabilitation program.Ventilatory efficiency will be calculated as the ratio of minute ventilation to carbon dioxide production.
Change from baseline in functional capacity. | From enrollment to the end of prehabilitation (15 sessions, 3 weeks).
  Change in functional capacity will be assessed using the one-minute-sit-to-stand test before and after the prehabilitation program. Performance during the one-minute-sit-to-stand test will be reported as the number of lifts during the test. The pre-specified minimal clinically important difference is set at 3 lifts.
Change from baseline in quadriceps muscle isometric strength. | From enrollment to the end of prehabilitation (15 sessions, 3 weeks).
  Change in maximum voluntary quadriceps muscle isometric strength will be assessed by dynamometry before and after the prehabilitation program. The pre-specified minimal clinically important difference is set at 7.5 Nm.
Change from baseline in inspiratory muscle strength. | From enrollment to the end of prehabilitation (15 sessions, 3 weeks).
  Change in inspiratory muscle strength will be assessed as maximal inspiratory pressure using manometry before and after the prehabilitation program. The pre-specified minimal clinically important difference is set at 13.5 cm H2O.
Change from baseline in expiratory muscle strength. | From enrollment to the end of prehabilitation (15 sessions, 3 weeks).
  Change in expiratory muscle strength will be assessed as maximal expiratory pressure using manometry before and after the prehabilitation program.
Change from baseline in peak expiratory flow. | From enrollment to the end of prehabilitation (15 sessions, 3 weeks).
  Change in peak expiratory flow will be assessed by flow meter during maximal expiratory effort before and after the prehabilitation program.
Change from baseline in peak cough expiratory flow. | From enrollment to the end of prehabilitation (15sessions, 3weeks).
  Change in peak cough expiratory flow will be assessed by flow meter during maximal cough effort before and after the prehabilitation program.
Change from baseline in quality of life. | From enrollment to the end of prehabilitation (15sessions, 3weeks).
  Change in quality of life will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-30) and its Lung Cancer module (LC 13) before and after the prehabilitation program. Scores range from 0 to 100 with a higher score reflecting either better function or milder symptoms. The pre-specified minimal clinically important difference is set at +3 points for improvement and -6 points for deterioration.
Change from baseline in symptoms of anxiety. | From enrollment to the end of prehabilitation (15sessions, 3weeks).
  Change in symptoms of anxiety will be assessed using the Hospital Anxiety and Depression questionnaire, anxiety subscore, before and after the prehabilitation program. The score ranges from 0 (best) to 21 (worst). The pre-specified minimal clinically important difference is set at -1.5 point.
Change from baseline in symptoms of depression. | From enrollment to the end of prehabilitation (15sessions, 3weeks).
  Change in symptoms of depression will be assessed using the Hospital Anxiety and Depression questionnaire, depression subscore, before and after the prehabilitation program. The score ranges from 0 (best) to 21 (worst). The pre-specified minimal clinically important difference is set at -1.5 point.
Adherence | At the end of prehabilitation (3 weeks).
  Adherence will be assessed as the ratio of completed sessions to prescribed sessions (15 sessions).
Post-operative complications. | Thirty days following surgery.
  Post-operative complications at 30 days following surgery will be assessed using the Clavien-Dindo classification. The pre-specified minimal clinically important difference between groups is set at 30%.
Clinically-relevant post-operative complications. | Thirty days following surgery.
  Post-operative complications at 30 days following surgery will be assessed using the Clavien-Dindo classification. Complications with a score equal or superior to two on this classification will be considered as clinically-relevant. The pre-specified minimal clinically important difference between groups is set at 30%.
Hospital length of stay following surgery | Thirty days following surgery.
  Hospital length of stay following surgery will be assessed as the number of days between surgery and discharge.
  Patient discharge is confirmed after validation of all the following items:
  Patient discharge is confirmed after validation of all the following items:
  * Patient is autonomous in eating, dressing, and toileting.
  * Autonomous in getting out of bed.
  * Autonomous in personal hygiene.
  * Autonomous in using the toilet.
  * Patient is able to walk 50 meters without desaturation below 90% (or return to -preoperative state).
  * Patient is able to climb and descend one flight of stairs without desaturation below 90% (or return to preoperative state).
  * Satisfactory wound healing.
  The pre-specified minimal clinically important difference is set at 1 day.
Environmental impact | At the end of prehabilitation (3 weeks).
  The environmental impact will be assessed using the Climate Partner Hub software (Climate Partner®, Munich, Germany). The assessment will include a Life Cycle Assessment for each device used in both groups, data transmission and storage on cloud servers for hybrid prehabilitation, and transportation for both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Bonnevie, PhD, Principal Investigator — Association ADIR; Fairuz Boujibar, PhD, Study Chair — Rouen University Hospital - Thoracic Surgery Department; Francis-Edouard Gravier, PhD, Study Chair — Association ADIR; Antoine Cuvelier, Prof, Study Chair — Association ADIR; Jean-François Muir, Prof, Study Chair — Association ADIR; David Debeaumont, MD, Study Chair — Rouen University Hospital - Department of Respiratory and Exercise Physiology; Jean-Marc Baste, Prof, Study Chair — Rouen University Hospital - Thoracic Surgery Department
Locations (1):
- Association ADIR, Rouen, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon reasonable request for research purposes after publication. This includes de-identified data related to demographic characteristics, as well as endpoints published either in the main manuscript or any supplemental data. Requests should be sent to t.bonnevie@adir-hautenormandie.com
Time Frame: Data will be made available after publication.
Access Criteria: Data will be made available upon request, for research purpose. Request should be send to t.bonnevie@adir-hautenormandie.com

REFERENCES:
- [Background] Gravier FE, Smondack P, Boujibar F, Prieur G, Medrinal C, Combret Y, Muir JF, Baste JM, Cuvelier A, Debeaumont D, Bonnevie T. Prehabilitation sessions can be provided more frequently in a shortened regimen with similar or better efficacy in people with non-small cell lung cancer: a randomised trial. J Physiother. 2022 Jan;68(1):43-50. doi: 10.1016/j.jphys.2021.12.010. Epub 2021 Dec 21. PMID 34952813